CLINICAL TRIAL: NCT00419822
Title: A Randomized, Intent to Treat, Controlled Study of the Efficacy of Verum Acupuncture Compared to Sham Acupuncture in the Management of Post Operative Symptoms in Breast Cancer Subjects That Have Undergone Axillary Surgery
Brief Title: Acupuncture in the Management of Post Operative Symptoms in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Legacy Health System (Other)
Responsible Party: Nathalie Johnson, MD, Legacy Health System
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCA-TCM-001
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2010-05

CONDITIONS: Breast Cancer
Keywords: Acupuncture; Range of Motion; Quality of Life
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Acupuncture (Active Comparator)
  Interventions: Procedure: Acupuncture
- Sham Acupuncture (Sham Comparator)
  Interventions: Procedure: Sham Acupuncture
- Standard of Care (Placebo Comparator)
  Interventions: Other: Patient to receive standard care without Acupuncture or Sham Acupuncture.

INTERVENTIONS:
Procedure: Acupuncture — 6 Acupuncture visits
  Arms: Acupuncture
Procedure: Sham Acupuncture — 6 Acupuncture visits with sham procedure
  Arms: Sham Acupuncture
Other: Patient to receive standard care without Acupuncture or Sham Acupuncture. — Standard care
  Arms: Standard of Care

SUMMARY:
This study is for the woman who will have axillary (armpit) surgery as part of their breast cancer treatment. The purpose of this project is to evaluate if acupuncture is helpful to control pain and improve range of motion (arm movement). Another goal is to find out if women have an improvement in their quality of life. This study is being done in collaboration with the Oregon College of Oriental Medicine (OCOM).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects
* Expected survival at least 6 months or greater
* Has had surgery with axillary dissection
* Greater than 6 nodes removed during surgery
* Greater than 21 years of age

Exclusion Criteria:

* Previous mastectomy
* Double mastectomy at the time of current axillary surgery
* Any diagnoses of autoimmune disease
* Pregnant or lactating women
* Unable to provide written informed consent
* Suspected or diagnosed fibromyalgia
* Previous shoulder injuries for the specific arm that will undergo axillary dissection
* Known or suspected drug or alcohol abuse as determined by the investigator
* Decreased range of motion (ROM) as evidenced on standard preoperative exam
* Previous acupuncture (lifetime)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-09; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Determine the difference in pain and range of motion | 3 months after surgery
Determine the difference in function | 3 months after surgery
Determine the difference in quality of life | 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Johnson, MD, Principal Investigator — Legacy Health System
Locations (1):
- Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon, United States

REFERENCES:
- See also: Related Info — http://www.legacyhealth.org